CLINICAL TRIAL: NCT04147858
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NYX-2925 in Subjects With Fibromyalgia
Brief Title: Efficacy and Safety of NYX-2925 in Subjects With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aptinyx (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NYX-2925-2005
Record Dates: First submitted 2019-10-29; First posted 2019-11-01 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — NYX-2925

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization algorithm, randomization allocation, allocation to study drug or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NYX-2925 50 mg (Experimental): NYX-2925 50 mg administered orally.
  Interventions: Drug: NYX-2925
- NYX-2925 100 mg (Experimental): NYX-2925 100 mg administered orally.
  Interventions: Drug: NYX-2925
- Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NYX-2925 — NYX-2925 administered orally
  Arms: NYX-2925 100 mg; NYX-2925 50 mg
Drug: Placebo — Placebo administered orally
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of NYX-2925 versus placebo for the treatment of fibromyalgia.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to assess the efficacy and safety of NYX-2925 in subjects with fibromyalgia.

This 13- to 16-week study will include a 1- to 4-week Screening Period followed by a 12-week double-blind, randomized, placebo-controlled Treatment Period.

ELIGIBILITY:
Inclusion criteria:

* Informed consent
* Subject has a history of fibromyalgia that was diagnosed >1 year prior to screening and reports at least moderate pain over the last week
* Stable protocol allowed medication and other therapies during the study
* Agrees to use highly effective birth control during the study
* Has not participated in an interventional study for at least 30 days and agrees not to participate in another interventional study during the study

Exclusion Criteria:

* Pain due to other conditions or diseases that would complicate participation in the study or pain reporting
* Current or historical serious medical conditions
* Prior participation in NYX-2925 clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Aptinyx Clinical Site, Phoenix, Arizona
  - Aptinyx Clinical Site, Culver City, California
  - Aptinyx Clinical Site, Fresno, California
  - Aptinyx Clinical Site, Orange, California
  - Aptinyx Clinical Site, Redlands, California
  - Aptinyx Clinical Site, Temecula, California
  - Aptinyx Clinical Site, Torrance, California
  - Aptinyx Clinical Site, Fernandina Beach, Florida
  - Aptinyx Clinical Site, Jacksonville, Florida
  - Aptinyx Clinical Site, Lady Lake, Florida
  - Aptinyx Clinical Site, Miami, Florida
  - Aptinyx Clinical Site, Orlando, Florida
  - Aptinyx Clinical Site, Palmetto Bay, Florida
  - Aptinyx Clinical Site, Winter Park, Florida
  - Aptinyx Clinical Site, Alpharetta, Georgia
  - Aptinyx Clinical Site, Chicago, Illinois
  - Aptinyx Clinical Site, Flossmoor, Illinois
  - Aptinyx Clinical Site, Gurnee, Illinois
  - Aptinyx Clinical Site, Skokie, Illinois
  - Aptinyx Clinical Site, Evansville, Indiana
  - Aptinyx Clinical Site, West Des Moines, Iowa
  - Aptinyx Clinical Site, Newton, Kansas
  - Aptinyx Clinical Site, Prairie Village, Kansas
  - Aptinyx Clinical Site, Wichita, Kansas
  - Aptinyx Clinical Site, Roslindale, Massachusetts
  - Aptinyx Clinical Site, Hazelwood, Missouri
  - Aptinyx Clinical Site, Omaha, Nebraska
  - Aptinyx Clinical Site, Las Vegas, Nevada
  - Aptinyx Clinical Site, Brooklyn, New York
  - Aptinyx Clinical Site, New York, New York
  - Aptinyx Clinical Site, Staten Island, New York
  - Aptinyx Clinical Site, Williamsville, New York
  - Aptinyx Clinical Site, Cincinnati, Ohio
  - Aptinyx Clinical Site, Oklahoma City, Oklahoma
  - Aptinyx Clinical Site, Duncansville, Pennsylvania
  - Aptinyx Clinical Site, Memphis, Tennessee
  - Aptinyx Clinical Site, Austin, Texas
  - Aptinyx Clinical Site, Houston, Texas
  - Aptinyx Clinical Site, Danville, Virginia
  - Aptinyx Clinical Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Started | 101 | 104 | 105 (One subject in the placebo group did not have post baseline efficacy measurements and is not included in efficacy results presented.)
Completed | 84 | 82 | 85
Not Completed | 17 | 22 | 20
Not completed — Adverse Event | 6 | 6 | 6
Not completed — Lack of Efficacy | 3 | 3 | 1
Not completed — Lost to Follow-up | 1 | 6 | 2
Not completed — Withdrawal by Subject | 3 | 4 | 10
Not completed — Subject Noncompliance, Other | 4 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- NYX-2925 50 mg: NYX-2925 50 mg administered orally once daily.
- NYX-2925 100 mg: NYX-2925 100 mg administered orally once daily.
- Placebo: Placebo administered orally once daily.
- Total: Total of all reporting groups
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo | Total
Number analyzed (Participants) | 101 | 104 | 105 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.81) | 51.8 (13.45) | 53.1 (12.28) | 52.7 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 99 | 96 | 289
  Male | 7 | 5 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 27 | 22 | 82
  Not Hispanic or Latino | 67 | 77 | 83 | 227
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 10 | 6 | 18 | 34
  White | 87 | 88 | 84 | 259
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 101 | 104 | 105 | 310

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Numerical Rating Scale (NRS) Score
Description: Change from baseline to Week 12 in the weekly mean of the daily Numerical Rating Scale (NRS) score assessing average pain intensity in the past 24 hours, scores range from 0-10, with higher scores indicating worse pain (0 being no pain and 10 being the worst possible pain)
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
units on a scale | -1.26 (1.603) | -1.47 (1.983) | -1.23 (1.846)
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 0.539, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 0.425, t-test, 2 sided

2. Secondary Outcome: Number of Subjects "Much Improved" or "Very Much Improved" on the Patient Global Impression of Change (PGI-C) at Week 12
Description: Number of subjects "much improved" or "very much improved" on the Patient Global Impression of Change (PGI-C) at Week 12
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
Participants | 22 | 24 | 24
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 0.824, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 1.000, t-test, 2 sided

3. Secondary Outcome: Daily Sleep Interference (DSIS) Score
Description: Change from baseline in the weekly mean of the Daily Sleep Interference Scale (DSIS) scores at Week 12; Response options range from 0 (Did not interfere with sleep) to 10 (Completely interfered with sleep, unable to sleep due to pain), with higher scores indicating greater interference with sleep.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
units on a scale | -1.42 (1.835) | -1.45 (2.104) | -1.38 (2.177)
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 0.297, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 0.603, t-test, 2 sided

4. Secondary Outcome: Number of Subjects Achieving ≥30% Pain Reduction
Description: Number of subjects achieving ≥30% reduction from baseline in the weekly mean NRS average pain intensity at Week 12; NRS Scores range from 0-10, with higher scores indicating worse pain (0 being no pain and 10 being the worst possible pain).
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
Participants | 30 | 34 | 29
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 0.871, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 0.352, t-test, 2 sided

5. Secondary Outcome: Number of Subjects Achieving ≥50% Pain Reduction
Description: Number of subjects achieving ≥50% reduction from baseline in the weekly mean NRS average pain intensity at Week 12; NRS scores range from 0-10, with higher scores indicating worse pain (0 being no pain and 10 being the worst possible pain)
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
Participants | 13 | 15 | 13
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 0.626, t-test, 2 sided

6. Secondary Outcome: Fibromyalgia Impact Questionnaire-Revised (FIQR) Score
Description: Change from baseline to Week 12 in the Fibromyalgia Impact Questionnaire - Revised (FIQR) score; FIQR scores range from 0-100, with higher scores indicating greater impact of fibromyalgia
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
units on a scale | -12.6 (20.10) | -12.3 (20.56) | -9.9 (20.08)
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 0.059, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 0.726, t-test, 2 sided

7. Secondary Outcome: Patient Reported Outcomes Measurement Information System - Fibromyalgia (PROMIS-FM) Sleep Disturbance Score
Description: Change from baseline to Week 12 in the PROMIS-FM sleep disturbance score, scores range from 0-40, with higher scores indicating greater sleep disturbance.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
units on a scale | -3.59 (8.238) | -3.93 (8.346) | -4.66 (9.567)
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 0.888, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 0.832, t-test, 2 sided

8. Secondary Outcome: Patient Reported Outcomes Measurement Information System - Fibromyalgia (PROMIS-FM) Fatigue Profile Score
Description: Change from baseline to Week 12 in the PROMIS-FM fatigue profile score, scores range from 0-80, with higher scores indicating greater impact of fatigue
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
units on a scale | -3.5 (8.70) | -3.7 (9.04) | -2.9 (7.90)
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 0.536, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 0.982, t-test, 2 sided

9. Secondary Outcome: Patient Reported Outcomes Measurement Information System - Fibromyalgia (PROMIS-FM) Physical Function Score
Description: Change from baseline to Week 12 in the PROMIS-FM physical function score, scores range from 0-60, with higher scores indicating greater difficulty with physical function.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
units on a scale | 2.18 (5.017) | 2.08 (5.223) | 1.83 (5.153)
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 0.190, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 0.764, t-test, 2 sided

10. Secondary Outcome: Use of Rescue Medication
Description: The number of subjects using rescue medication.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 104
Participants | 93 | 87 | 88
Statistical Analysis 1: Comparison: NYX-2925 50 mg vs Placebo; Test type: Superiority; p = 0.097, t-test, 2 sided
Statistical Analysis 2: Comparison: NYX-2925 100 mg vs Placebo; Test type: Superiority; p = 0.849, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are defined as the start of the event occurring on or after the date of first dispensed study drug (Day 1, Baseline Visit) and before or on the last dose (Week 12). The protocol required adverse events to be followed to resolution of the adverse event.
Description: MedDRA (24.1)
Arm/Group | NYX-2925 50 mg | NYX-2925 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/104 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/101 | 2/104 | 0/105
Other Adverse Events (participants affected / at risk) | 18/101 | 19/104 | 18/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NYX-2925 50 mg (N=101) | NYX-2925 100 mg (N=104) | Placebo (N=105)
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NYX-2925 50 mg (N=101) | NYX-2925 100 mg (N=104) | Placebo (N=105)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 9 (11)
Fatigue (General disorders) | 3 (3) | 1 (1) | 3 (4)
COVID-19 (Infections and infestations) | 2 (2) | 6 (6) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 6 (7) | 2 (2)
Headache (Nervous system disorders) | 8 (8) | 4 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT04147858/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT04147858/SAP_001.pdf